CLINICAL TRIAL: NCT01908673
Title: Automatic Self Transcending Meditation (ASTM) Versus Heart Rate Variability (HRV) Biofeedback in Patients With Late Life Depression (LLD): a Randomized Controlled Longitudinal Pilot Feasibility Study
Brief Title: Automatic Self Transcending Meditation (ASTM) Versus Heart Rate Variability (HRV) Biofeedback in Patients With Late Life Depression (LLD): a Longitudinal Pilot Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSREB 103966
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Late Life Depression
Keywords: heart rate variability biofeedback; automatic self transcedental meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HRV biofeedback (Active Comparator): heart rate variability biofeedback
  Interventions: Behavioral: HRV biofeedback
- ASTM (Active Comparator): Automatic Self Transcedental Meditation
  Interventions: Behavioral: ASTM

INTERVENTIONS:
Behavioral: HRV biofeedback
  Arms: HRV biofeedback
Behavioral: ASTM
  Other Names: Automatic Self Transcedental Meditation
  Arms: ASTM

SUMMARY:
Background: Depression in the elderly, also known as late life depression (LLD) is common and its prevalence ranges from 2 to 6% in the community. Heart Rate Variability (HRV), a physiological autonomic variable is reduced in LLD and this might have implications for cardiovascular events including death. Methods to improve HRV in LLD have not been adequately assessed. Automatic Self-Transcending Meditation (ASTM) is a simple yet powerful technique that allows the mind to become calm and peaceful. HRV biofeedback is a method of teaching individuals to voluntarily improve HRV and other physiological functions to a prescribed range.This pilot study attempts to investigate feasibility of these interventions and provide preliminary data regarding the effectiveness of these techniques.

Hypothesis: ASTM and HRV biofeedback are feasible and their effectiveness for improving HRV in patients with LLD can be assessed.

Methods: Participants with LLD between the ages of 66 and 80 will be randomized to either ASTM or HRV biofeedback after optimizing them on antidepressant therapy. Participants will receive training and continue practice in either of these techniques over a period of twelve weeks. HRV and secondary measures will be assessed pre and post at the end of study period.

Expected Results and Significance: The investigators expect to find both techniques to be feasible treatments for those with LLD. Results from this pilot study will help to assess the potential for successful implementation of a future larger study which will evaluate the efficacy of these treatments for improving HRV.

ELIGIBILITY:
Inclusion Criteria:

1. Of either gender, age 66-80 years.
2. Have an Axis 1 diagnosis of major depressive disorder (DSM IV code 296.2x or 296.3x) (comorbid anxiety and dysthymic disorder will be acceptable).
3. HAMD-24 score of >20.
4. Low risk of suicide as elicited by clinical interview.
5. Being able to sit for 30-45 minutes, without physical pain
6. Of general good physical health with no severe cardiovascular disease in the past 12 months (myocardial infarction, stroke or TIA).
7. No past history of neurological disease or seizures.
8. Sufficient hearing to comprehend verbal instructions without the need to lip read.
9. Able to attend regular outpatient follow-up appointments.

Exclusion Criteria:

1. Incapable of giving informed consent to study participation.
2. Participating in other similar studies.
3. Other significant Axis I diagnosis (including PTSD, OCD, Panic Disorder, Bipolar Affective Disorder, Substance dependence, Dementia)
4. Psychotic episodes within the past 12 months.
5. Recent (within the past 6 months) head trauma that required emergency care
6. Currently on an antidepressant from the classes of Tricyclic antidepressants, Monoamine oxidase (MAO) inhibitors, or Serotonin Noradrenaline Reuptake inhibitors (SNRI) such as venlafaxine, desvenlafaxine or duloxetine.
7. Currently practicing any type of formal meditation, mindfulness or breathing techniques.
8. Mini Mental Score Exam (MMSE) ≤18

Ages: 66 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) | Week 0 and week 12
  HRV will be assessed at baseline and at end of study period (week 12)

SECONDARY OUTCOMES:
Change in depression severity | week 0 and week 12
  Depression symptoms will be assessed on the Hamilton depression rating scale (HAM-D, 24 items), Clinical Global Impression (CGI), and self-rated Geriatric Depression Scale (GDS)

CONTACTS AND LOCATIONS:
Overall Officials: Akshya Vasudev, MBBS MD MRCPSych, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada